CLINICAL TRIAL: NCT02360306
Title: The Analysis of the EBUS Scope as a Hybrid Bronchoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Lonny Yarmus, Assistant Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00081049
Record Dates: First submitted 2014-11-07; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Lymphadenopathy
MeSH Terms: conditions — Lymphadenopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional EBUS (Active Comparator): Subjects in this arm will have endobronchial ultrasound bronchoscopy done by the conventional EBUS scope rather than the hybrid EBUS scope. Subjects in this arm, like in the Hybrid EBUS arm, may or may not receive transbronchial forcep biopsies, airway brusings, and/or radial EBUS, depending on clinical need.
  Interventions: Procedure: Endobronchial Ultrasound
- Hybrid EBUS (Experimental): Subjects in this arm will have endobronchial ultrasound bronchoscopy done by the hybrid EBUS scope rather than the conventional EBUS scope. Subjects in this arm, like in the conventional EBUS arm, may or may not receive transbronchial forcep biopsies, airway brusings, and/or radial EBUS, depending on clinical need.
  Interventions: Procedure: Endobronchial Ultrasound

INTERVENTIONS:
Procedure: Endobronchial Ultrasound — Endobronchial ultrasound bronchoscopy with potential transbronchial needle aspiration, transbronchial forcep biopsy, brushing, or radial endobronchial ultrasound

SUMMARY:
Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is widely used in the diagnosis of mediastinal and hilar adenopathy as well as in staging in lung cancer patients. Many studies have confirmed the utility of EBUS-TBNA with high sensitivity, specificity, and accuracy for the diagnosis of mediastinal and hilar adenopathy. 1-3 Less well reported has been the use of the EBUS bronchoscope to perform other procedures such as transbronchial biopsy (TBBx), endobronchial biopsy (EBBx), bronchoalveolar lavage (BAL) and airway brushings. While not well reported in the medical literature, anecdotal evidence supports these practices. The investigators propose a methodological evaluation of the full spectrum of procedures that have been performed and that are possible using an EBUS bronchoscope.

DETAILED DESCRIPTION:
1. Objectives (include all primary and secondary objectives)

   Primary objective - To study and more fully describe the full spectrum of procedures performed using an EBUS bronchoscope outside of EBUS-TBNA.
2. Background (briefly describe pre-clinical and clinical data, current experience with procedures, drug or device, and any other relevant information to justify the research)

   There currently exists only anecdotal evidence and individual reports of the use of EBUS bronchoscopes in the performance of non-EBUS-TBNA procedures. Given the full size working channel through which all standard bronchoscopic tools are able to pass, the EBUS bronchoscope has been reported to have been used in the performance of other procedures such as BAL, TBBx, EBBx and airway brushing. Frequently during bronchoscopic procedures in which EBUS-TBNA is used to sample lymph nodes within the hilum and mediastinum there exists a need to perform other procedures including but not limited to those listed above. In these cases, the EBUS bronchoscope is removed and exchanged for a standard video bronchoscope often times dirtying the scope for only a single procedure. We routinely use EBUS bronchoscopy in our daily practice as interventional pulmonologists and would like to study the use of these bronchoscopes in the performance of procedures other than TBNA perhaps in an effort to more fully understand the benefits and limitations associated with the use of an EBUS bronchoscope during conventional video bronchoscopy.
3. Study Procedures

   1. Study design

      We plan to collect the data for all clinically indicated procedures using an EBUS bronchoscope over a twelve month time frame in the JHH outpatient endoscopy suite. No procedures will be performed for research purposes. No additional procedures will be performed outside the scope of standard practice.
   2. Study duration and number of study visits required of research participants. 12 month study duration, no research visits will be required.
   3. Justification of why participants will not receive routine care or will have current therapy stopped.

      All patients will receive routine standard of care.
   4. Justification for inclusion of a placebo or non-treatment group. The study is aimed at analyzing the data generated by clinically indicated procedures thus no placebo or non-treatment group has been included in the study.
4. Drugs/ Substances/ Devices

   a. The rationale for choosing the drug and dose or for choosing the device to be used.

   The rationale for studying the EBUS bronchoscope and its application to non-TBNA procedures is to study the actual use of the scopes as well as to ascertain whether an EBUS scope is able to perform all bronchoscopic procedures thus decreasing the need for extra bronchoscopes and decreasing cleaning costs and wear on the devices.
5. Benefits a. Description of the probable benefits for the participant and for society. There will be no direct benefit to the participants but society may benefit the medical society if EBUS bronchoscopes are shown to be able to perform the full range of bronchoscopic procedures as there may be decreased costs to the medical system as well as potential reduction in procedure time by eliminating the need to exchange scopes mid procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing bronchoscopy involving the use of an EBUS bronchoscope in the Johns Hopkins endoscopy suite over the course of the study period

Exclusion Criteria:

* Patients not able to safely undergo bronchoscopy as judged by the Interventional Pulmonary service and Anesthesia. This follows standard clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Procedures able to be performed succesfully by Hybrid EBUS | twelve months
  Procedures able to be performed succesfully by Hybrid EBUS in comparison to Conventional EBUS. This will be assessed using a case report form that includes a checklist of various procedures (e.g. TBNA, transbronchial forcep biopsy)

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States